CLINICAL TRIAL: NCT06529692
Title: Mi-SPA: Michigan Split-belt Adaptation Paradigm to Improve Knee Loading After Anterior Cruciate Ligament Reconstruction (Aim 3)
Brief Title: Michigan Split-belt Treadmill Training Program to Improve Long-Term Knee Biomechanics After ACL Reconstruction
Acronym: Mi-SPA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Riann Palmieri-Smith, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00221406_Aim3; 1R21AR082643 (NIH)
Record Dates: First submitted 2024-07-26; First posted 2024-07-31 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: ACL; Anterior Cruciate Ligament; ACL Injury
Keywords: Biomechanics; Knee Loading; Split-Belt Treadmill; Asymmetric Walking
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Early Stance Training (Experimental): This study arm will complete 6-weeks of a split-belt treadmill training program. The program will require participants to walk on a split-belt treadmill 2 times a week for 20 minutes with the ACL leg walking at 150-170% of 1.1 m/s and the Non-ACL leg walking at 1.1 m/s.
  Interventions: Behavioral: Split-Belt Training
- Mid-Stance Training (Experimental): This study arm will complete 6-weeks of a split-belt treadmill training program. The program will require participants to walk on a split-belt treadmill 2 times a week for 20 minutes with the ACL leg walking at 30-50% of 1.1 m/s and the Non-ACL leg walking at 1.1 m/s.
  Interventions: Behavioral: Split-Belt Training
- Placebo Split-Belt Training (Placebo Comparator): This study arm will complete 6-weeks of a split-belt treadmill training program. The program will require participants to walk on a split-belt treadmill 2 times a week for 20 minutes with the ACL leg walking at a speed that is 10% different from 1.1 m/s and the Non-ACL leg walking at 1.1 m/s.
  Interventions: Behavioral: Placebo Split-Belt Training

INTERVENTIONS:
Behavioral: Placebo Split-Belt Training — Walking on a split-belt treadmill in which the belt under the ACL leg will move at a speed that is minimally slower than the other belt.
  Arms: Placebo Split-Belt Training
Behavioral: Split-Belt Training — Walking on a split-belt treadmill in which the treadmill belt under the ACL leg will move at a speed faster or slower than the belt under the Non-ACL leg.
  Arms: Early Stance Training; Mid-Stance Training

SUMMARY:
The goal of this study is to gather pilot data to help inform a future clinical trial. As such, the investigators will employ a randomized clinical trial design, but data will only be collected on 9 total subjects. Nine subjects will be randomized to 2 split-belt intervention groups (one group where early stance loading is trained and the other where midstance loading is trained) and a placebo group.

The goal of this study is to explore the adaptations in knee loading from a 6-week split-belt training intervention.

The investigators' main question for this aim is:

1. Does knee loading, measured by the sagittal plane knee moment, change to a greater extent in the split-belt treadmill training groups compared to the placebo group?
2. Are there differences in training-related knee loading changes between individuals trained in the early stance vs. midstance loading split-belt training?

DETAILED DESCRIPTION:
It is commonplace for individuals after anterior cruciate ligament (ACL) reconstruction to shift mechanical demands away from their surgical knee and limb. This manifests as diminished knee moments and vertical ground reaction forces in the ACL limb during everyday tasks (e.g., walking, running, standing, landing, etc.) and persists for as long as 2.5 years after surgery. This pattern of underloading is considered maladaptive, as it has been linked to re-injury and biological markers that are consistent with the development of post-traumatic osteoarthritis that affects over 50% of knees 10-20 years after surgical reconstruction.

Split-belt treadmill training is a gait retraining approach where treadmill belt speeds are decoupled (i.e., one belt is set to move at a faster or slower speed than the other belt) during walking. Split-belt training is based on well-established motor learning principles, such as error-based learning and variability of practice which can lead to locomotor adaptations. In healthy individuals, split-belt treadmill walking significantly increases (from baseline) knee moment impulses in the limb on the slow belt than on the fast belt during the braking and propulsive phases of gait. Split-belt treadmill training has also shown promise in individuals with neurological deficits, resulting in significant improvements in gait biomechanics after training.

To explore the adaptations in loading from a 6-week split-belt training intervention, the investigators will conduct a pilot randomized clinical trial design, but data will only be collected on 9 total subjects. Nine subjects will be randomized to one of 3 groups: 1) early stance split-belt treadmill training, 2) mid-stance split-belt treadmill training, or 3) placebo split-belt treadmill training. The primary outcome, sagittal plane knee moment, will be examined before, midway, & after the 6-weeks of training. Other outcomes, vertical ground reaction force, knee joint contact force, and the Knee Injury and Osteoarthritis Outcome Score, will be measured at the same timepoints. Medial and lateral knee cartilage thickness are additional outcomes that will only be assessed before and after training.

ELIGIBILITY:
Inclusion Criteria:

* aged 14-45 years
* suffered an acute, complete ACL rupture as confirmed by MRI and physical exam
* have undergone ACL reconstruction w autograft within the past 10 months
* willingness to participate in testing and follow-up as outlined in the protocol
* English-speaking

Exclusion Criteria:

* inability to provide written informed consent
* female subjects who are pregnant or are planning to become pregnant (self-reported)
* previous ACL injury
* previous surgery to either knee
* bony fracture accompanying ACL injury
* patients who experienced a knee dislocation
* patients who had their ACL reconstructed with an allograft
* patients who underwent a multi-ligamentous and/or staged ACL reconstruction

Ages: 14 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-08-13 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
ACL Leg Sagittal Plane Knee Moment | Before training, midway through training (3 weeks), & after training (6 weeks)
  Peak Sagittal Plane Knee Moment recorded during walking gait

OTHER OUTCOMES:
Non-ACL Leg Sagittal Plane Knee Moment | Before Training, midway through training (3 weeks), & after training (6 weeks)
  Peak Sagittal Plane Knee Moment recorded from the Non-ACL leg during walking gait
ACL Leg Vertical Ground Reaction Force | Before Training, midway through training (3 weeks), & after training (6 weeks)
  Peak Vertical Ground Reaction Force recorded from the ACL leg during walking gait
Non-ACL Leg Vertical Ground Reaction Force | Before Training, midway through training (3 weeks), & after training (6 weeks)
  Peak Vertical Ground Reaction Force recorded from the Non-ACL leg during walking gait
ACL Leg Internal Knee Joint Contact Force | Before Training, midway through training (3 weeks), & after training (6 weeks)
  Internal knee joint reaction force for the ACL limb estimated using musculoskeletal modeling
Non-ACL Leg Internal Knee Joint Contact Force | Before Training, midway through training (3 weeks), & after training (6 weeks)
  Internal knee joint reaction force for the Non-ACL limb estimated using musculoskeletal modeling
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Before Training, midway through training (3 weeks), & after training (6 weeks)
  The KOOS score is a percentage from 0-100, with 0 representing extreme knee problems and 100 representing no knee problems. A higher score indicates fewer knee issues, while a lower score indicates more.
Medial Cartilage Thickness | Before (0 weeks) & after training (6 weeks)
  Thickness of the cartilage from the medial femoral trochlea measured using ultrasound
Lateral Cartilage Thickness | Before (0 weeks) & after training (6 weeks)
  Thickness of the cartilage from the lateral femoral trochlea measured using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Riann M Palmieri-Smith, PhD, ATC, Principal Investigator — University of Michigan; Chandramouli Krishnan, PT, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made publicly available via Deep Blue Data which is managed by the University of Michigan.
Supporting Information: Study Protocol, ICF
Time Frame: We will strive to release data to the repository as rapidly as it is possible to analyze experiments and publish results. Data used in publications will be released at the time of publication.